CLINICAL TRIAL: NCT06479239
Title: Phase I/II Study of Anti-CD3 x Anti-EGFR Bispecific Antibody (EGFRBi) Armed Fresh Peripheral Blood Mononuclear Cells (EGFR FPBMC) in Metastatic or Unresectable Pancreatic Cancer
Brief Title: Study of EGFRBi Armed Fresh PBMC in Metastatic or Unresectable Pancreatic Cancer
Acronym: Panc 002
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Tri Minh Le, MD, Associate Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR231503
Record Dates: First submitted 2024-06-17; First posted 2024-06-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Pancreas Cancer; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EGFR Fresh Peripheral Blood Mononuclear Cells (Experimental): Participants will undergo apheresis to collect cells to make EGFR fresh peripheral blood mononuclear cells (FPBMC). These cells will be activated in the lab to fight against pancreas cancer. About 3-4 days after apheresis, participants will start receiving infusions of EGFR FPBMC. Throughout treatment, participants will have blood taken for labs, to check disease status and also to look at immune response. Study treatment will stop if the participant has disease progression. Participants that have disease progression after the first 8 infusions may receive chemotherapy and then continue study treatment with the other 8 infusions.
  Interventions: Drug: EGFR FPBMC

INTERVENTIONS:
Drug: EGFR FPBMC — Participants will receive 8 weekly infusions of EGFR FPBMC, then 8 additional infusions every 2 weeks.

SUMMARY:
The purpose of this study is to understand the safety and estimate the efficacy of combining anti-cluster of differentiation 3 (CD3) x anti-Epidermal Growth Factor Receptor (EGFR) bispecific antibody fresh peripheral blood mononuclear cells (EGFR FPBMC) for patients with metastatic or unresectable pancreas cancer. Participants receive 8 weekly doses and then 8 more doses every 2 weeks of EGFR FPBMC by intravenous infusion.

DETAILED DESCRIPTION:
Once subjects are determined to be eligible, white blood cells (lymphocytes) are collected via leukapheresis procedure. The T cells in the mononuclear cells are coated with bispecific antibody to activate the T cells and the mononuclear cells are reinfused into the patients so the T cells can multiply and kill tumors.

About 72 hours after the leukapheresis procedure, EGFR FPBMC infusions will start. After about 8-9 weeks, participants will have another leukapheresis procedure and then receive doses every 2 weeks for 8 more doses. Before, throughout and following EGFR FPBMC, research blood will be collected to better understand immune response. Disease status will be checked regularly during and after study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed locally advanced pancreatic cancer (LAPC)/unresectable pancreatic cancer (UPC) or metastatic pancreatic cancer (MPC) not eligible for curative intent therapy
2. Received at least 1 line of chemotherapy and have stable disease (SD) or better for 3 months prior to enrollment. Therapy should consist of either a gemcitabine, 5FU-based (including capecitabine) or albumin-bound paclitaxel-based regimen. Patients with actionable mutations should have received targeted therapy prior to enrollment on trial. Patients who qualify for immunotherapy due to mismatch repair protein/microsatellite stable and tumor mutational burden status should also have received immunotherapy prior to enrollment on trial.
3. Measurable disease by immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
5. Age ≥ 18 years
6. Females of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment/registration
7. Females of childbearing potential and males must agree to use an effective method for contraception for the duration of the treatment with study drug plus 90 days (duration of sperm turnover). Males must also abstain from sperm donations during study treatment and for at least 90 days after the last dose of study drug.
8. Adequate organ function within 14 days prior to registration, defined as the following:

   * Absolute neutrophil count >= 500/mm3
   * Absolute lymphocyte count >= 400/mm3
   * Platelets >= 75,000/mm3
   * Hemoglobin >= 8 g/dL
   * Serum creatinine < 2.0mg/dL or calculated/measured creatinine clearance >= 50 ml/min
   * Bilirubin <= 2 mg/dL
   * Aspartate transferase (AST) and Alanine transaminase (ALT) <= 5.0 x upper limit of normal (ULN)
   * Alpha gal < 0.35 IU/ml or "negative"
9. Ability to provide informed consent and provision of written informed consent
10. Stated willingness to comply with all study procedures and availability for the duration of the study
11. Adequate cardiac function as defined as:

    * No uncontrolled angina or severe ventricular arrhythmias
    * No clinically significant pericardial disease
    * No history of myocardial infarction (MI) in the last year before registration
    * No Class 3 or higher New York Heart Association Congestive Heart Failure

Exclusion Criteria:

1. Known hypersensitivity to cetuximab
2. Treatment with investigational agent within 3 weeks prior to registration
3. Serious non-healing wound, ulcer, bone fracture, major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration
4. Known active liver disease, human immunodeficiency virus (HIV)+ or evidence of active Hepatitis C or B virus; bleeding or condition associated with high-risk bleeding (anticoagulation is allowed)
5. Active infection; prior antibiotic/antifungal/antiviral therapies within 2 weeks prior to registration
6. History of a myocardial infarction within 1 year prior to registration
7. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
8. Autoimmune disease that has required systemic treatment with chronic steroids or immunosuppressive therapy in the 2 years prior to registration (thyroxine, insulin, or corticosteroid replacement is allowed)
9. History or evidence of any condition that might confound the results of the trial, interfere with the subject's participation, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
10. Females must not be currently breast feeding.
11. The treating investigator feels the patient is not able to be compliant.
12. History of active Bacillus Tuberculosis (TB).
13. Has received a live vaccine within 30 days of registration.
14. Prisoners or patients who are incarcerated.
15. Patients who are compulsorily detained for treatment of a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) during the dose escalation phase (during the first 8 infusions only) | Through the dose escalation phase (during the first 8 infusions only, about 8 weeks after starting study treatment))
  As defined in the protocol

SECONDARY OUTCOMES:
Overall Response Rate | Through the dose escalation phase (during the first 8 infusions only, about 8 weeks after starting study treatment))
  Number/Percentage of participants that have a partial or complete response to study treatment
Progression free survival | Through 3 years after last infusion for each participant (a maximum of about 3 1/2 years)
  Time from start of treatment to time of progression or death from any cause, whichever occurs first.
Overall Survival | Through 3 years after last infusion for each participant (a maximum of about 3 1/2 years)
  Time from start of treatment to time of death from any cause.
Specific cytotoxicity by PBMCs against pancreatic cancer cell lines | Before study treatment, about 8-9 weeks into study treatment, then 30-45 days, 6 months and 12 months after completion of study treatment
  In blood samples
Development of antibodies to pancreatic cancer antigens | Before study treatment, about 8-9 weeks into study treatment, then 30-45 days, 6 months and 12 months after completion of study treatment
  In blood samples
Survival of EGFR FPBMCs after multiple infusions | Prior to study treatment, prior to each of the first 5 infusions, (optionally) about 1-2 days after each of the first 8 infusions, and about 8-10 weeks after starting study treatment
  In blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Tri Le, MD, DSc, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No